CLINICAL TRIAL: NCT00410137
Title: Influence of Nutritional and Inflammational Status on Survival of Hemodialysis Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Other Study IDs: 43/06
Record Dates: First submitted 2006-12-10; First posted 2006-12-12 (Estimated); Last update posted 2006-12-12 (Estimated); Status verified 2006-12

CONDITIONS: Inflammation; Body Composition
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
prospective longitudinal measurements of nutritional status parameters (body composition by BIA, anthropometry and biochemical indexes), inflammatory response (CRP, inflammatory cytokines (IL-1, IL-6, IL-10),IGF-1, leptin and NOx blood levels) and morbidity and mortality data collection over 2 year period in patients receiving chronic hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age > 18 years, in chronic hemodialysis treatment at least 3 months
* Stable and adequate hemodialysis treatment three months prior to participation in study as defined by Kt/V > 1.2 and/or hemodialysis performed 4 hours 3 times weekly
* Patients with normal hydration status (edema-free), with no neuro-muscular diseases
* Informed consent obtained before any trial-related activities

Exclusion Criteria:

* Patients with edema, pleural effusion or ascites at their initial assessment
* Patients with active malignant disease or liver cirrhosis
* Patients with neuro-muscular diseases
* Patients on chronic treatment with steroids on doses > 10 mg/day Prednisone (or equivalent)
* Patients treated with immunosuppressive agents
* Patients suffering from

  * Acute vasculitis
  * Severe systemic infections
  * Heart failure (NYHA class III-IV)
* The receipt of any investigational drug within 1 month prior to initiating of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-03; Study Completion 2008-04

CONTACTS AND LOCATIONS:
Overall Officials: Ilia Beberashvili, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf-Harofeh Medical Center, Ẕerifin, Israel